CLINICAL TRIAL: NCT00228280
Title: Periapical Bone Healing After Apicectomy With and Without Retrograde Root Filling
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Professor, Ann Wenzel, department of Oral Radiology, School of Dentistry, University of Aarhus, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: journal n. 20050041
Record Dates: First submitted 2005-09-23; First posted 2005-09-28 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Stomatognathic Disease; Mouth Disease; Periapical Disease; Alveolar Bone Loss
Keywords: Apicoectomy; Retrograde; MTA
MeSH Terms: conditions — Stomatognathic Diseases; Mouth Diseases; Periapical Diseases; Alveolar Bone Loss | interventions — mineral trioxide aggregate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Mineral Trioxide Aggregate (MTA) — retrograde rootfilling with MTA or smoothening of the orthograde root-filling, gutta-percha
  Other Names: retrograde root filling material; retrofilling

SUMMARY:
Ph.D project: Periapical bone healing after apicectomy with and without retrograde root filling.

The aim of this study is to assess periapical bone healing after apicectomy without a filling and apicectomy combined with a retrograde filling material, MTA. Further, we will estimate risk factors in non-healing cases.

Study hypothesis: There is no difference in treatment outcome between:

Periapical bone healing after apicectomy with retrograde root filling and Periapical bone healing after apicectomy without retrograde root filling

DETAILED DESCRIPTION:
Ph.D project: Periapical bone healing after apicectomy with and without retrograde root filling.

60 patients have been selected from a group of 490 patients, who had a full mouth radiographic status taken in connection with a population study of apical periodontitis in Aarhus Community. The selection criteria for the 60 patients were patients with a persisting apical periodontitis, Periapical Index (PAI) score 3-5, on front teeth and premolars in the upper jaw. The orthograde root filling in the tooth must be at least 2 years old and sufficient regarding density and length.

The 60 patients will be randomised into the two groups of apicectomy with and without filling. A radiograph will be taken just before the operation and 6 and 12 months after the operation. In the assessment of bone healing, we will use two different techniques, subtraction radiography and the Periapical Index (PAI).

We will also evaluate the benefits of using the operation microscope during the operation, and if clinical photos can be useful as documentation of treatment result.

ELIGIBILITY:
Inclusion Criteria:

healthy person age 18 or above sufficient root filling sufficient coronal restauration apical infection for at least 2 years Pai Score3, 4, or 5

Exclusion Criteria:

boneless more than 50 % communication between pocket and apical infection no visible root filling material after apicectomy facial bone less than 3 mm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-01; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Periapical bone healing Pai score | one-year

SECONDARY OUTCOMES:
Periapical bone healing bone density | one-year

CONTACTS AND LOCATIONS:
Overall Officials: Ann Wenzel, professor, Study Director — faculty of health science, royal dental collegue, department of Oral Radiology, Aarhus
Locations (1):
- Faculty of Health Science, Aarhus, Aarhus C, Denmark

REFERENCES:
- See also: Department of Oral Radiology, Royal Dental Colleague, Aarhus, Denmark — http://www.odont.au.dk/rad/default.html